CLINICAL TRIAL: NCT00460694
Title: A Phase II Trial on Allogeneic Cytokine-induced Killer Cell Immunotherapy for Relapse After Allogeneic Marrow Transplant for Haematological Malignancies
Brief Title: Allogeneic Cytokine-induced Killer Immunotherapy for Relapse After Allogeneic Marrow Transplant for Haematological Malignancies
Acronym: alloCIK
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIK#2/2007; NMRC/1097/2006
Record Dates: First submitted 2007-04-12; First posted 2007-04-16 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Chronic Myeloid Leukemia; Non Hodgkin's Lymphoma; Hodgkin's Disease; Myelodysplastic Syndrome; Multiple Myeloma
Keywords: allogeneic transplant; haematological malignancies; allogeneic CIK cells
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Lymphoma, Non-Hodgkin; Hodgkin Disease; Myelodysplastic Syndromes; Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: infusion of allogeneic CIK cells — infusion of allogeneic CIK cells at graded doses

SUMMARY:
Cytokine-induced killer ( CIK ) cells have been shown by our lab to be cytolytic against both autologous and allogeneic acute myeloid leukemia ( AML ) cells. Large scale expansion of CIK cells has also been shown to be feasible in healthy allogeneic stem cell donors as well as in patients undergoing mobilization for autologous transplant.

Donor lymphocyte infusion (DLI) has been shown to be active against some haematological malignancies including CML, AML, MDS,NHL and Hodgkin's disease. These donor lymphocytes can be further activated in vitro to become CIK cells. At least 2 other centers in the world have given allogeneic CIK cells for patients relapsing post allogeneic transplant for a variety of haematological malignancies. These early reports have demonstrated feasibility, absence of increased GVHD and possible efficacy in some cases.

We are proposing a Phase I /II study on the feasibility / efficacy of immunotherapy with allogeneic CIK cells for patients who relapse after allogeneic marrow transplant for their haematological malignancies. These patients have to be either refractory to conventional donor lymphocyte infusion, or need a larger number of donor lymphocyte than could be provided by unmanipulated donor lymphocytes. Donor lymphocytes will be collected and cultured in GMP facilities to maturity, then infused into patients. This will be given in graded doses at 4 weekly intervals and continued on in the absence of GVHD till remission is achieved or disease progression occurs. Patients may receive various forms of chemotherapy appropriate to the clinical condition in each case before the allogeneic CIK infusion.

Efficacy will be assessed by comparing the response to allogeneic CIK infusion vs that to due to conventional DLI, ie response to the two different treatment using DLI response as the comparator. We expect about 10 such cases to be done over the next 3 years. Significant statistics is unlikely to be generated but observation and description of the response can generate useful information for presence or not of the efficacy of such a treatment.

If clinical efficacy and superiority over conventional DLI is demonstrated, then future allogeneic CIK may take the place of DLI in this group of poor prognosis patients who relapse after allogeneic transplant .

DETAILED DESCRIPTION:
1. Patient inclusion criteria This trial includes only patients who have relapsed after an allogeneic transplant, who have either 1.1 No response to conventional DLI given for at least one dose, or 1.2 No possibility of access to large number of donor lymphocyte for repeated doses of DLI, This applies to cases of unrelated transplant or cord blood transplant

   1,3 Patients who developed significant GVHD to conventional DLI, but had no other therapeutic option. In such cases the rationale is based on mice studies of mismatched CIK producing much less GVHD than mismatched unmanipulated splenocytes.
2. Collection of peripheral blood stem cells ( PBSC ) Sibling allogeneic donors will routinely have their PBSC harvested for the purpose of infusion into the recipients. Currently our practice involves one additional day of collection to freeze as backup to be used for DLI in the event of relapse. This collection is frozen in a few aliquots, and is available for CIK culture when need arises

   For cord blood transplant, one issue is that DLI is not available. There is one report on growing CIK from residual cells in the bags of cord blood after infusion, then stored frozen for use in future if need arises. This does not in anyway compromise the cord blood infusion. Similarly this can be done in the case of unrelated donor transplant. This will serve as a backup in the event that donor is not available for repeat collection of lymphocyte.
3. Culture of CIK cells

For culture from frozen product, this is rapidly thawed and culture started in gas permeable bags in complete medium and cytokine as detailed in SOP attached ( appendix 1 ). Culture medium and cytokine are added periodically till maturation of CIK at between 21-28 days.

For culture from residual cells in the thawed cord blood infusion bags, cells may need to undergo ficoll to remove rbc, then start culture in the similar way

3. Harvesting of CIK cells

At maturity between D21-D28, all bags of CIK cells are pooled and washed using COBE 2991 cell harvester. This will ensure removal of >99.9% of the original culture medium. Cells are then frozen and aliquots sent for quality control to ensure compliance to GMP standard. This includes bacteriological and fungal culture, mycoplasma and endotoxin testing.

4. Infusion of CIK cells Patients may undergo cytoreductive chemotherapy or oral immunosuppressive therapy as deemed fit in each individual case by the attending physician. At the nadir of lymphopenia , CIK cells are rapidly thawed at bedside and infused.

Dose and schedule of CIK cells follows the following principle 4.1 First dose for patients who have already received DLI and showed resistance : at double or triple the last DLI dose ( expressed as CD3/kg ).

4.2 First dose for patients who have not received any DLI : this will follow the conventional practice of DLI where the first dose will be 10 million CD3/kg.

4.3 Subsequent doses will be given at 4-weekly intervals allowing time to observe for development of GVHD and response.

4.3.1 If no response was observed, dose will be doubled or tripled ( depending on the size of the available aliquot ). If there is good response, dose will remain the same as the previous infusion.

4.3.2 In the presence of GVHD, infusion will be withheld till resolution of GVHD, then resumed at half or one-third of the previous dose ( depending on the size of the available aliquot).

4.4 Duration of CIK infusion will depending on the response status 4.4.1 In responding patients, 4-weekly CIK infusion will continue till a complete remission is achieved and then another 2-3 infusions beyond.

4.4.2 In patients who achieve a stable partial response, CIK infusion will continue in a 4-weekly interval, provided no adverse effect and CIK cells are available. This will continue on and stop if disease breaks through.

4.4.3 In patients where disease continues to progress after 2-3 cycles of CIK infusion, no further infusion will be given

ELIGIBILITY:
Inclusion Criteria:

This trial includes only patients who have relapsed after an allogeneic transplant, who have either:

1. No response to conventional DLI given for at least one dose, or
2. No possibility of access to large number of donor lymphocyte for repeated doses of DLI, This applies to cases of unrelated transplant or cord blood transplant
3. Patients who developed significant GVHD to conventional DLI, but had no other therapeutic option. In such cases the rationale is based on mice studies of mismatched CIK producing much less GVHD than mismatched unmanipulated splenocytes.

In view of the period taken to culture the cell to maturity, patient must have a life expectancy of more than one month. Interim measures eg chemotherapy or conventional DLI will be given during the interval so that ongoing treatment will not be compromised in any way.

Exclusion Criteria:

1. Uncontrolled infection or significant bleeding
2. Unstable vital signs
3. Any degree of hypoxia requiring oxygen therapy.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2006-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Feasibility of expansion of frozen donor mononuclear cells into CIK | 2 year
Toxicity including GVHD and marrow aplasia | 1 year from infusion for each patient

SECONDARY OUTCOMES:
Efficacy in terms of disease response as compared to previous treatment modality ie unmanipulated DLI | 2 years from infusion for each patient

CONTACTS AND LOCATIONS:
Overall Officials: Yeh-Ching Linn, MBBS, MRCP, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

REFERENCES:
- [Background] 1. YC Linn, LC Lau, KM Hui Generation of cytokine-induced killer cells from leukemic samples with in vitro cytotoxicity against autologous and allogeneic leukemic blasts British Journal of Haematology, 2002, 116: 78-86 2. C Sheffold, M Edinger, R S Negrin A Phase I trial of autologous cytokine-indueced killer cells for transplant of relapsed Hodgkin's disease and Non Hodgkin's lymphoma Biol of Blood and Marrow Transplant 2005, 11:181-187 3. Hao Jiang, Kaiyan Liu, Chunrong Tong, Bin Jiang, Daopei Lu The efficacy of chemotherapy in combination with autologous cytokine-induced killer cellsi n acute leukemia Chinese J Internal Med 2005, 44(3): 198-201 4. Jeanette Baker, Michael R Vernais, Maki Ito et al Expansion of cytolytic CD8+ natural killer T cells with limited capacity for graft-versus- host disease induction due to interferon gamma productin Blood, 2001, 97(!)(: 2923-2931 5. Ginna G Laport, Kevin Sheehan, Robert Lowsky et al Cytokine Induced Killer (CIK) cells as post transplant immunotherapy following allogeneic haemopoietic cell transplantation (Oral session ) Blood 2006, 108 (11) #412 6.Martino Introna, Gianmaria Borleri, Elena Conti et al Infusion of donor derived Cytokine-induced Killer Cells may induce clinical remission with limited GVHD in patients relapsing after allogeneic stem cell transplantation ( poster session) Blood 2006, 108(11), #3698 7. David L Porter, Bruce L Levine, Nancy Bunin et al A phase I trial of donor lymphocyte infusions expanded and activated ex vivo via CD3/CD28 costimulation Blood 2006, 107 (4), 1325-1331